CLINICAL TRIAL: NCT00365807
Title: Effectiveness of a Treatment Program for Pediatric Obesity
Brief Title: Examination of a Treatment Program for Overweight Children, Adolescents, and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R40MC06631-01-00
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Behavioral treatment; Family involvement
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Family Intervention (Primarily education) (Active Comparator): Behaviorally based family group intervention using standard education and nutrition counseling. Three hours of client contact
  Interventions: Other: Brief Family Intervention (Primarily education)
- Positively Fit (Experimental): 12 week (90 minute per session) behavioral group intervention for children and their parents. Children and parent attend parallel group with identical (but developmentally appropriate) information presented.
  Interventions: Behavioral: Positively Fit

INTERVENTIONS:
Behavioral: Positively Fit — 12-week group intervention for children with obesity and their parents/caregivers
  Arms: Positively Fit
Other: Brief Family Intervention (Primarily education) — 3 hours of contact with registered dietician for education and nutritional counseling.
  Arms: Brief Family Intervention (Primarily education)

SUMMARY:
The current study examined the effectiveness of a behaviorally-based group intervention for overweight children and their families. The target intervention was compared to an enhanced standard of care treatment. The impact of both treatment programs on numerous outcomes was explored.

DETAILED DESCRIPTION:
The primary objective of the present investigation was to determine the effectiveness of an empirically supported intervention for pediatric overweight in two outpatient clinical settings. A number of previous randomized clinical trials have demonstrated the efficacy of behaviorally-based group interventions for overweight children and their families. As called for by Kazdin and Weisz (1998) and Chambless and Hollon (1998) the proposed investigation was designed to demonstrate the effectiveness of such a treatment in a clinical setting, and to examine the effects of the intervention on children's quality of life (QOL). Because the clinical impact of empirically supported interventions is mitigated by economic and consumer variables, a secondary aim of the proposed investigation was to examine (1) the cost-effectiveness of an outpatient group intervention for pediatric obesity, and (2) the consumer satisfaction with the proposed intervention. Finally, an additional exploratory aim was to examine predictors of adherence to treatment for the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child between ages 7 and 17 (inclusive)
* Child BMI at or above the 85th percentile based on norms provided for age and gender
* Child's parent/guardian provides informed consent for treatment of the child as well as consent for study participation
* Child's parent/caregiver is willing to participate with the child in the program

Exclusion Criteria:

* Presence of serious mental illnesses or significant developmental delay that would reasonably predict altered ability to adhere to the treatment protocol
* Current physical illness or hospitalization of the child that would interfere with group attendance or protocol adherence

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2006-07; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
BMI Percentile Change | Treatment completion, 1 year follow up

SECONDARY OUTCOMES:
Quality of Life - The PedsQL™ (version 4.0;Varni et al., 2001) | treatment completion, one year follow up
Child Psychosocial Adjustment -- the Behavioral Assessment System for Children- Parent report form (BASC-PRF) and the BASC-Child Self Report (BASC-CSR; Reynolds & Kamphaus, 2002) | Treatment completion, one year follow up
Cost-effectiveness | Treatment completion, one year follow up
Consumer Satisfaction | Treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Ric G Steele, Ph.D., Principal Investigator — University of Kansas; Ann M. Davis, Ph.D., Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas, Lawrence, Kansas

REFERENCES:
- [Result] Steele RG, Aylward BS, Jensen CD, Cushing CC, Davis AM, Bovaird JA. Comparison of a family-based group intervention for youths with obesity to a brief individual family intervention: a practical clinical trial of positively fit. J Pediatr Psychol. 2012 Jan-Feb;37(1):53-63. doi: 10.1093/jpepsy/jsr057. Epub 2011 Aug 18. PMID 21852343